CLINICAL TRIAL: NCT00084396
Title: A Phase 2 Trial Of 4 Months Preoperative Letrozole 2.5 mg Daily For Postmenopausal Women With Estrogen Receptor Positive And/Or Progesterone Receptor Positive T2, T3, T4a-c, N0-2, M0 Breast Cancer- Novel Biomarkers for Aromatase Inhibitor Therapy
Brief Title: Neoadjuvant Letrozole in Treating Postmenopausal Women With Estrogen-Receptor Positive and/or Progesterone-Receptor Positive Stage II, Stage IIIA, or Stage IIIB Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000361963; R01CA095614 (NIH); P30CA091842 (NIH); WU-03-0586; UCSF-02755; UCSF-H8409-21398-04
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Letrozole/Surgery (Experimental)
  Interventions: Drug: letrozole; Procedure: conventional surgery

INTERVENTIONS:
Drug: letrozole
Procedure: conventional surgery

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using letrozole may fight breast cancer by reducing the production of estrogen. Giving letrozole before surgery may shrink the tumor so that it can be removed.

PURPOSE: This phase II trial is studying how well neoadjuvant letrozole works in treating postmenopausal women who are undergoing surgery for estrogen-receptor positive or progesterone-receptor positive stage II, stage IIIA, or stage IIIB breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Develop a predictive model of response (based on gene expression profiling) in postmenopausal women with estrogen- and/or progesterone-receptor positive stage II, IIIA, or IIIB breast cancer treated with neoadjuvant letrozole.

Secondary

* Determine the response rate in patients treated with this drug.
* Determine changes in Ki67 proliferation rates in patients treated with this drug.
* Determine the rate of improvement in surgical outcomes in patients treated with this drug.
* Determine the long-term outcomes in patients treated with this drug.
* Determine the safety of this drug in these patients.
* Determine mechanisms of resistance to this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive neoadjuvant oral letrozole once daily for 16 weeks in the absence of disease progression. Patients then undergo breast surgery one day after the last dose of letrozole. Patients with partial response after 16 weeks may continue to receive letrozole for an additional 8 weeks before undergoing breast surgery.

Patients are followed within 4 weeks after definitive surgery and then annually for 10 years.

PROJECTED ACCRUAL: A total of 150 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed infiltrating adenocarcinoma of the breast by core needle biopsy

  * Clinical stage T2-T4a-c, N0-2, M0
* Palpable and measurable disease
* Previously untreated disease
* Benefits from neoadjuvant therapy that would improve surgical outcome AND meets criteria for 1 of the following:

  * Marginal candidate for lumpectomy (e.g., lumpectomy feasible but patient at risk for positive margins or poor cosmetic outcome) AND patient desires breast-conserving surgery
  * Ineligible for lumpectomy due to size of primary tumor, but modified radical mastectomy feasible AND patient desires breast-conserving surgery
  * Inoperable disease AND systemic therapy required for disease to become operable by modified radical mastectomy
* Bilateral primary tumors allowed provided both tumors are consistent with entry criteria
* No inflammatory carcinoma (defined as peau d' orange affecting at least one third of the breast)

  * Direct extension of the tumor to the skin allowed
* No metastatic breast disease, except isolated ipsilateral supraclavicular lymphadenopathy
* Hormone receptor status:

  * Estrogen- and/or progesterone-receptor positive disease based on 10% or more nuclear staining of the invasive component of the tumor

PATIENT CHARACTERISTICS:

Age

* Postmenopausal

Sex

* Female

Menopausal status

* Postmenopausal, defined as meeting 1 of the following criteria:

  * Cessation of menstrual periods for at least 1 year
  * Bilateral surgical oophorectomy
  * Follicle-stimulating hormone and estradiol levels in the postmenopausal range

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* No severe liver dysfunction that would preclude study participation

Renal

* Not specified

Other

* Willing and able to provide biopsy material
* Willing to undergo breast surgery after neoadjuvant treatment
* No condition (e.g., confusion, infirmity, or alcoholism) that would preclude study compliance
* No other concurrent active and progressive invasive malignancies
* No other concurrent severe disease that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy or biological response modifiers for breast cancer

Chemotherapy

* No prior chemotherapy for breast cancer
* No concurrent chemotherapy for breast cancer

Endocrine therapy

* At least 2 weeks since prior hormone replacement therapy or phytoestrogenic herbal, alternative, or over-the-counter (OTC) sex hormone remedies
* No prior hormonal agents for breast cancer
* No prior aromatase inhibitors, tamoxifen, raloxifene, or other antiestrogen or selective estrogen receptor modulators
* No concurrent drugs known to affect sex hormone status, including hormone replacement therapy or phytoestrogenic herbal, alternative, or OTC remedies
* No other concurrent endocrine therapy for breast cancer

Radiotherapy

* No prior radiotherapy for breast cancer
* No concurrent radiotherapy for breast cancer

Surgery

* Prior sentinel node biopsy allowed
* No other concurrent surgery for breast cancer

Other

* More than 30 days since prior non-approved or experimental drugs
* Concurrent bisphosphonates for osteoporosis allowed
* No other concurrent treatment for breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2003-10; Primary Completion 2007-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Predictive model for response as assessed by gene expression profiling

SECONDARY OUTCOMES:
Response rate
Changes in Ki67 proliferation rates
Rate of improvement in surgical outcomes
Long-term outcomes
Safety
Mechanisms of resistance

CONTACTS AND LOCATIONS:
Overall Officials: Michael Naughton, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States